CLINICAL TRIAL: NCT06136520
Title: The Effect of Baby Massage Training Given to Pregnant Women on Maternal Attachment and Postpartum Depression: A Randomized Controlled Study
Brief Title: The Effect of Baby Massage Training Given to Pregnant Women on Maternal Attachment and Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/132
Record Dates: First submitted 2023-10-26; First posted 2023-11-18 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-04

CONDITIONS: Baby Massage; Postpartum Depression
Keywords: Postpartum Depression; baby massage; attachment
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After the first measurements are made and the groups are determined; "Personal Information Form", "Perinatal Attachment Inventory" and "Beck Depression Inventory" will be applied to the experimental and control groups. Pregnant women in the experimental group were 32-40 weeks of pregnancy.
  After baby massage training is given, 30-42 weeks after birth. between days and 60-72. "Maternal Attachment Scale" and "Edinburgh Postpartum Depression Scale" will be applied to the experimental and control groups on the following days. The control group will receive standard care while the experimental group receives training. After the second postpartum data of the pregnant women in the control group are collected, a 30-minute baby massage training will be given by the researcher.
  Interventions: Behavioral: Baby massage
- Control group (No Intervention): The control group will receive standard care while the experimental group receives training. After the second postpartum data of the pregnant women in the control group are collected, a 30-minute baby massage training will be given by the researcher.

INTERVENTIONS:
Behavioral: Baby massage — After the first measurements are made and the groups are determined; "Personal Information Form", "Perinatal Attachment Inventory" and "Beck Depression Inventory" will be applied to the experimental and control groups. Pregnant women in the experimental group were 32-40 weeks of pregnancy.
  After baby massage training is given, 30-42 weeks after birth. between days and 60-72. "Maternal Attachment Scale" and "Edinburgh Postpartum Depression Scale" will be applied to the experimental and control groups on the following days. The control group will receive standard care while the experimental group receives training. After the second postpartum data of the pregnant women in the control group are collected, a 30-minute baby massage training will be given by the researcher.
  Arms: experimental group

SUMMARY:
The research to be conducted within the scope of the project will be randomized controlled, and the population of the research will be primiparous pregnant women reached through social media. Primiparous pregnant women in the 32nd - 40th weeks of pregnancy will be included in the study, and the sample size is determined by using the G*Power (3.1.9.2) program, considering a margin of error of 0.05 and data loss, with a power of 95% and a medium effect size; 27 people should be included in the experimental (baby massage) group and 27 people in the control group. In determining the groups, participants will be assigned to experimental and control groups using the "Randomizer.org" program. Pregnant women included in the research will be informed about the study and will be presented with an "Informed Consent Form" and "Voluntary Consent Form". Baby massage training will be given to the experimental group, and a reminder training will be given 2 weeks later. "Personal Information Form", "Prenatal Attachment Inventory" and "Beck Depression Inventory" will be applied to both groups at the beginning of the study, and postpartum 30-42 weeks. and 60-72. "Maternal Attachment Scale" and "Edinburg Postpartum Depression Scale" will be administered between days.

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 18-35, Being primiparous and having a singleton pregnancy,

* No high-risk pregnancy,
* Being in the 32nd to 40th week of pregnancy,
* Being literate and knowing and understanding Turkish,
* Pregnant women who have internet access and knowledge of internet usage.

Exclusion Criteria:

* ● Presence of chronic disease,

  * Pregnancy with congenital malformation,
  * Unwanted pregnancy,
  * Having attended a pregnancy school,
  * Women who become pregnant as a result of assisted reproductive technology,
  * Those with hearing and vision problems,
  * Having a known serious psychiatric disease diagnosis.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
the Maternal Attachment Scale (mother-baby bonding scale) | 3 months
  Postpartum ages 30-42 in the Maternal Attachment Scale "Experimental Group". days and 60-72. It will be applied to mothers between days. Postpartum ages 30-42 are in the "Control Group" of the Maternal Attachment Scale. days and 60-72. It will be applied to mothers between days.
  Measures maternal feelings and behaviors that show love The lowest score obtained from the scale is 26, the highest score is 104, and a high score indicates high maternal attachment.
The Edinburgh Postpartum Depression Scale | 3 months
  The Edinburgh Postpartum Depression Scale will be used to evaluate and monitor the postpartum depression development levels of the groups. The cut-off score of the scale is 12/13, and women who score above 13 are considered to be at risk for depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Betül Uncu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No